CLINICAL TRIAL: NCT00377897
Title: Optimisation d'un Produit de thérapie Cellulaire Autologue Par Cellules mononucléées médullaires Dans l'ischémie Critique Des Membres inférieurs liée à l'athérosclérose
Brief Title: Cell Therapy With Bone Marrow Mononuclear Cells in Critical Leg Ischemia (CLI)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Paris 5 - Rene Descartes (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: DRC, APHP
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPTIPEC
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Critical Leg Ischemia
Keywords: critical leg ischemia; PAD; cell therapy
MeSH Terms: interventions — Cell- and Tissue-Based Therapy

INTERVENTIONS:
Procedure: cell therapy — Injection of Bone-Marrow mononuclear cells in the muscles of the calf.

SUMMARY:
This study will treat by cell therapy 20 patients with critical leg ischemia (CLI) not eligible for revascularization or angioplasty. It will use exactly the same protocol as published by Tateishi-Yuyama et al. (Lancet 2002), using bone-marrow mononuclear cells (BMMNC).

DETAILED DESCRIPTION:
Patients will be included with CLI according to the TASC criteria. Under general anesthesia, 500 ml of bone marrow is harvested in both iliac crests. After isolation and concentration of the BMMNC in 30 ml, 40 injections of around 0.75 ml will be done in the gastrocnemius of the ischemic leg, within 3 hours after preparation of the cell therapy product.

Patients will then be followed-up every week during one month and then every month during one year.

This study was approved by the ethical committee of Paris-Broussais HEGP (France) and our french regulatory agency (AFSSAPS).

It began including patients in January 2005 and will last until December 2007.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Signature of informed consent
* Critical leg ischemia with ankle pressure < 70 mmHg
* Ischemic ulcer or gangrene
* No possibility of surgical revascularization
* No possibility of angioplasty

Exclusion Criteria:

* Cancer
* Suspicion of a cancer on X-Ray, mammography or elevated PSA
* Age < 18
* Life expectancy < 6 months
* Active retinopathy
* Angioplasty or surgical revascularization within 3 months
* Stoke within 3 months
* HIV + or HCV/HBC+

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-01; Primary Completion 2008-09 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Ankle brachial index | 6 months
Healing | 1 year
Amputation rate | 1 year

SECONDARY OUTCOMES:
TcPO2 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Emmerich, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Emmerich, Paris, Paris, France

REFERENCES:
- [Derived] HoWangYin KY, Loinard C, Bakker W, Guerin CL, Vilar J, d'Audigier C, Mauge L, Bruneval P, Emmerich J, Levy BI, Pouyssegur J, Smadja DM, Silvestre JS. HIF-prolyl hydroxylase 2 inhibition enhances the efficiency of mesenchymal stem cell-based therapies for the treatment of critical limb ischemia. Stem Cells. 2014 Jan;32(1):231-43. doi: 10.1002/stem.1540. PMID 24105925
- [Derived] Smadja DM, Duong-van-Huyen JP, Dal Cortivo L, Blanchard A, Bruneval P, Emmerich J, Gaussem P. Early endothelial progenitor cells in bone marrow are a biomarker of cell therapy success in patients with critical limb ischemia. Cytotherapy. 2012 Feb;14(2):232-9. doi: 10.3109/14653249.2011.627917. Epub 2011 Oct 31. PMID 22040109
- [Derived] Smadja DM, d'Audigier C, Guerin CL, Mauge L, Dizier B, Silvestre JS, Dal Cortivo L, Gaussem P, Emmerich J. Angiogenic potential of BM MSCs derived from patients with critical leg ischemia. Bone Marrow Transplant. 2012 Jul;47(7):997-1000. doi: 10.1038/bmt.2011.196. Epub 2011 Oct 10. No abstract available. PMID 21986637
- [Derived] Smadja DM, d'Audigier C, Bieche I, Evrard S, Mauge L, Dias JV, Labreuche J, Laurendeau I, Marsac B, Dizier B, Wagner-Ballon O, Boisson-Vidal C, Morandi V, Duong-Van-Huyen JP, Bruneval P, Dignat-George F, Emmerich J, Gaussem P. Thrombospondin-1 is a plasmatic marker of peripheral arterial disease that modulates endothelial progenitor cell angiogenic properties. Arterioscler Thromb Vasc Biol. 2011 Mar;31(3):551-9. doi: 10.1161/ATVBAHA.110.220624. Epub 2010 Dec 9. PMID 21148423